CLINICAL TRIAL: NCT00135590
Title: Evaluation of the Effectiveness of a Protein Pulse-Feeding Pattern in Elderly Patients
Acronym: PRO-PULSé
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PO30418; AOR03003
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2004-11

CONDITIONS: Protein-Energy Malnutrition
Keywords: Protein pulse-feeding; Nutritional supplementation; Protein-energy malnutrition; Elderly subjects; Body composition
MeSH Terms: conditions — Protein-Energy Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Protein pulse-feeding
  Interventions: Dietary Supplement: Protein pulse-feeding
- 2 (Active Comparator): Spread diet
  Interventions: Dietary Supplement: Spread diet

INTERVENTIONS:
Dietary Supplement: Protein pulse-feeding — Dietary protein (80% of daily intake) was consumed in one meal (12.00h)
  Arms: 1
Dietary Supplement: Spread diet — Dietary protein was spread over the four meals.
  Arms: 2

SUMMARY:
The researchers tested the hypothesis that a protein pulse-feeding pattern was more efficient in improving muscle mass and immune functions than was a protein spread-feeding pattern, after 45 days, in elderly malnourished patients.

DETAILED DESCRIPTION:
To estimate the amelioration of the accretion in protein and the immunizing deficit thanks to a nutrition "PULSEE" ( to hold on 80 % of the proteic by day in on meal) with a proteic distributed all along the day for old subjects having a denutrition

To also estimate that the diminution of the morbidity decrease (infections, bedsores) the average during the stay and the mortality according to 2 modalities of grip nutritional

ELIGIBILITY:
Inclusion Criteria:

* Must be malnourished
* Hospitalization into a geriatric rehabilitation care unit
* Age > 70 years
* C-reactive protein (CRP) < 50 mg/l

Exclusion Criteria:

* Enteral or parenteral nutrition
* Renal, cardiac or digestive insufficiency
* Diabetes
* Pacemaker
* Mini-Mental State (MMS) < 15

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Lean mass (dual energy X-ray absorptiometry [DEXA] and bioelectrical-impedance analysis [BIA]) | 42 days

SECONDARY OUTCOMES:
Immune functions | 42 days
Hand-grip strength | 42 days
Biological nutritional parameters | 42 days
Mortality and morbidity (infections and bedsores) | 42 days
Activity of Daily Living (ADL) | 42 days
Plasmatic amino acid levels | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Aussel Christian, PHD, PharmD, Study Director — Assistance Publique Hopitaux de Paris:Laboratoire de Biologie de la Nutrition EA 2498 and Hôpital Emile Roux (AP-HP); Cynober Luc, PHD, PharmD, Study Chair — Assistance Publique Hopitaux de Paris:Laboratoire de Biologie de la Nutrition EA 2498 and Hôpital Hôtel-Dieu (AP-HP); Bouillanne Olivier, MD, Principal Investigator — Assistance Publique Hopitaux de Paris:Laboratoire de Biologie de la Nutrition EA 2498 and Hôpital Emile-Roux (AP-HP)
Locations (1):
- Hôpital Emile-Roux (AP-HP), Limeil-Brévannes, France

REFERENCES:
- [Derived] Bouillanne O, Neveux N, Nicolis I, Curis E, Cynober L, Aussel C. Long-lasting improved amino acid bioavailability associated with protein pulse feeding in hospitalized elderly patients: a randomized controlled trial. Nutrition. 2014 May;30(5):544-50. doi: 10.1016/j.nut.2013.10.006. Epub 2013 Oct 14. PMID 24355438
- [Derived] Bouillanne O, Curis E, Hamon-Vilcot B, Nicolis I, Chretien P, Schauer N, Vincent JP, Cynober L, Aussel C. Impact of protein pulse feeding on lean mass in malnourished and at-risk hospitalized elderly patients: a randomized controlled trial. Clin Nutr. 2013 Apr;32(2):186-92. doi: 10.1016/j.clnu.2012.08.015. Epub 2012 Aug 30. PMID 22992307